CLINICAL TRIAL: NCT04616417
Title: Investigational Oocyte Cryopreservation for Medical and Non Medical Indications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Sana Salih, Principal Investigator, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012-0233
Record Dates: First submitted 2020-10-30; First posted 2020-11-05 (Actual); Results first posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-02

CONDITIONS: Infertility, Female; Deferred Childbearing
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Investigational Oocyte Cryopreservation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational Oocyte Cryopreservation (Experimental): All subjects will undergo controlled ovarian hyperstimulation. They will be treated with variable dosages of injectable gonadotrophins over a period of 8 to 12 days. Response will be monitored using vaginal ultrasound and serum estradiol levels. When appropriate follicle maturation has been achieved, a single dose of human chorionic gonadotropin (hCG) will be administered to induce final oocyte maturation. Thirty-six hours after hCG administration, the subject will undergo standard transvaginal oocyte retrieval under ultrasound guidance. The procedure takes approximately 20 minutes and is carried out under conscious sedation with Fentanyl and Versed. The oocytes are immediately handed off to the embryology technicians in the IVF laboratory.
  Interventions: Procedure: Investigational Oocyte Cryopreservation

INTERVENTIONS:
Procedure: Investigational Oocyte Cryopreservation — Transvaginal oocyte retrieval under ultrasound guidance

SUMMARY:
This is a prospective study to assess the long term benefits and outcomes of the existing oocyte cryopreservation methods for fertility preservation in women with a potential medical or non medical risk of loss of fertility

DETAILED DESCRIPTION:
This is a prospective study to assess the long term benefits and outcomes of the existing oocyte cryopreservation methods for fertility preservation in women with a potential medical or non medical risk of loss of fertility. Women wishing to preserve their oocytes using cryopreservation will be informed of the risk and limitations of the procedures involved in ovarian hyperstimulation, oocyte recovery, cryopreservation and subsequent viability after warming. Women who consent to the procedure will undergo standard controlled ovarian hyperstimulation (COH) and oocyte retrieval procedures currently in use for IVF. Following harvest all eggs obtained will be evaluated for degree of fragmentation and maturation status. The oocytes will be cryopreserved using kits of media and devices currently approved for use in the vitrification of fertilized eggs and embryos, and the cryopreserved oocytes will be stored for future patient use in a long term storage facility in Minnesota (Reprotech Ltd.). Patients with stored oocytes will be contacted annually to determine the outcome of any oocyte warming procedures (oocyte thawing, fertilization and embryo transfer).

We will obtain a structured fertility focused quality of life questionnaire (FertiQol) and survey to assess one year after harvest the impact of the process. We will compare medical (cancer) patients to those patients undergoing oocyte cryopreservation for non-medical reasons

ELIGIBILITY:
Inclusion Criteria:

* Women aged >18 and < 40years
* Women able to defer definitive cancer therapy for 21 to 30 days
* Women diagnosed with cancer or any disease whose treatment or its progression may impair their reproductive potential (this would include but not be limited to cancer patients requiring treatment with chemotherapy or radiation, patients with rheumatologic diseases such as lupus, rheumatoid arthritis and ulcerative colitis and patients with genetic predisposition to cancers
* Women undergoing standard In Vitro Fertilization to treat infertility who experience unforeseen events that halts the treatment cycle
* Women seeking oocyte cryopreservation for non medical reasons, such as deferred childbearing
* Women who are carriers of BRCA mutations predisposing them to cancer
* Otherwise healthy females
* Ability and willingness to comply with study protocol
* Informed written consent, prior to any study-related procedure not part of normal care, with the understanding that the subject may withdraw consent at any time without prejudice to their future medical care

Exclusion Criteria:

* Current pregnancy
* Serum FSH > 10 mIU/ml for patients having egg freezing for a medical indication
* Serum FSH > 10 mIU/ml for patients having egg freezing for social reasons
* Women with psychological, psychiatric, or other conditions which prevent giving fully informed consent (Post Traumatic Stress Disorder, severe depression, bipolar disorder, schizophrenia, severe anxiety and inability to cope)
* Patients with extensive disease whose therapy is deemed palliative by the medical oncologist

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 29 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sana Salih, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Hospital & Health Sciences System - IVF Program in the Fertility Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Oocyte Cryopreservation
Started | 29
Cancer Patients Who Completed Follow up Interview and Fertility Qulaity of Life Questionnaire | 1
Patients With Non-medical Reasons Who Completed Interview Fertility Quality of Life Questionnaire | 9
Completed | 20
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Oocyte Cryopreservation
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Fertility Quality of Life Questionnaire Completed After One Year After Oocyte Cryopreservation for Non-medical Reasons
Description: We will obtain a structured fertility focused quality of life questionnaire (FertiQol) and survey to assess one year after harvest the impact of the process. We will compare cancer patients to those patients undergoing oocyte cryopreservation for non-medical reasons. FertiQol is scored based on the standards of the assessment tool in a quantitative manner. Only 9 patients completed the this questionnaire. FertiQoL consists of 36 items that assess core (24 items) and treatment-related (10 items) quality of life as well as overall life and physical health (2 items). Higher scores indicated better outcomes and lower scores indicated worse outcomes on this questionnaire.
Time Frame: Fertility quality of life questionnaire completed after one year after oocyte cryopreservation
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Oocyte Cryopreservation
Number analyzed (Participants) | 9
Participants | 9

2. Primary Outcome: Structured Clinical Interview Completed After One Year After Oocyte Cryopreservation for Non-medical Reasons
Description: Study participants will be contacted on an annual basis using the "Investigational Oocyte Cropreservation Follow-up Call Script/structured interview" to determine any subsequent attempts to utilize the stored oocytes for the purpose of initiating a pregnancy, along with the outcome of the attempt. Only 9 patients completed this interview. There was not score assigned to this interview.
Time Frame: structured clinical interview completed after one year after oocyte cryopreservation
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Oocyte Cryopreservation
Number analyzed (Participants) | 9
Participants | 9

3. Primary Outcome: Fertility Quality of Life Questionnaire Completed After One Year After Oocyte Cryopreservation for Cancer Patients
Description: We will obtain a structured fertility focused quality of life questionnaire (FertiQol) and survey to assess one year after harvest the impact of the process. We will compare cancer patients to those patients undergoing oocyte cryopreservation for non-medical reasons. FertiQol is scored based on the standards of the assessment tool in a quantitative manner. only one cancer patient completed this questionnaire.FertiQoL consists of 36 items that assess core (24 items) and treatment-related (10 items) quality of life as well as overall life and physical health (2 items). Higher scores indicated better outcomes and lower scores indicated worse outcomes on this questionnaire.
Time Frame: Fertility Quality of Life Questionnaire Completed After One Year After Oocyte Cryopreservation for cancer patients
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Oocyte Cryopreservation
Number analyzed (Participants) | 1
Participants | 1

4. Primary Outcome: Structured Clinical Interview Completed After One Year After Oocyte Cryopreservation for Cancer Patients
Description: study participants will be contacted on an annual basis using the "Investigational Oocyte Cropreservation Follow-up Call Script/structured interview" to determine any subsequent attempts to utilize the stored oocytes for the purpose of initiating a pregnancy, along with the outcome of the attempt. only 1 cancer patient completed this structured interview. There was not score assigned to this interview.
Time Frame: Structured Clinical Interview Completed After One Year After Oocyte Cryopreservation for cancer patients
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Oocyte Cryopreservation
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Investigational Oocyte Cryopreservation
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2022-03-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT04616417/Prot_000.pdf